CLINICAL TRIAL: NCT04118933
Title: An Exploratory Study for PD-1 Antibody JS001 in Participants With Microsatellite Instability-high (MSI-H) Advanced or Recurrent Colorectal Cancer
Brief Title: A Study for PD-1 Antibody JS001 in MSI-H Advanced or Recurrent Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xu jianmin (Other)
Responsible Party: Sponsor-Investigator, Xu jianmin, Deputy director of the colorectal cancer center, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K19406-JS001-ISS-141
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MSI-H advanced colorectal cancer (Experimental)
  Interventions: Drug: JS001

INTERVENTIONS:
Drug: JS001 — JS001 240mg, Q3W

SUMMARY:
To observe the efficacy of PD-1 antibody JS001 in the treatment of participants with microsatellite instability-high (MSI-H) advanced or recurrent colorectal cancer, so as to provide sufficient evidence for MSI-H as a biomarker of PD-1/PD-L1 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and sign informed consent voluntarily;
* Histologically confirmed advanced or recurrent colorectal cancer, and MSI detection identified MSI-H;
* Patients who have previously received first-line or above chemotherapy or targeted therapy and failed to the treatment or experienced recurrence;
* At least one measurable lesion (RECIST 1.1);
* Agree to provide tumor tissue samples and Pathology reports related to the specimens;
* Aged 18 to 75 years, gender not limited;
* Eastern Cooperative Oncology Group(ECOG) performance status(PS) 0-1; 8. Expected survival ≥3 months;
* Laboratory test values must meet the following standards within 7 days before enrollment;
* Women of reproductive age must confirm that the serum pregnancy test is negative and agree to use effective contraceptive measures during the study drug use

Exclusion Criteria:

* Uncontrolled or symptomatic hypercalcemia;
* Had major surgery or had not fully recovered from previous surgery within 4 weeks before enrollment;
* central nervous system(CNS) metastases;
* Bone metastases;
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (once a month or more frequently) allow the patient to have a catheter indwelling;
* Having a history of idiopathic pulmonary fibrosis, organic pneumonia;
* Uncontrolled active infection, including but not limited to acute pneumonia;
* Have other malignant tumors at the same time;
* The patient has any active autoimmune diseases or a history of autoimmune diseases;
* Liver diseases of known clinical significance, including active viral viral hepatitis, alcoholic hepatitis or other hepatitis, cirrhosis, fatty liver and hereditary liver diseases.
* Previous use of anti-PD-1 antibody, anti-PD-l1 antibody, anti-PD-l2 antibody or anti-CTLA-4 antibody;
* Patients with active tuberculosis (TB);
* Received systemic immunosuppressive within 4 weeks prior to day 1 of the first cycle;
* Pregnancy test positive;
* Known human immunodeficiency virus (HIV) infection;
* A history of severe allergy, anaphylaxis or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins;
* Those who are known to be allergic to biological drugs produced by hamster ovary cells in China, or to citric acid monohydrate, sodium citrate dihydrate, mannitol and polysorbate (components of the experimental drugs);
* Patients who have previously received allogeneic stem cells or parenchymal organ transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2020-07-17 (Estimated); Study Completion 2021-07-17 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 12 Weeks from the drug firstly being taken
  The 12 week objective response will be measured according to RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China